CLINICAL TRIAL: NCT04104568
Title: Effectiveness of an Online Training and Support Program (iSupport Portuguese Version) to Reduce Burden, Depression and Anxiety and to Improve Quality of Life, Positive Aspects of Caregiving and Self-efficacy in Informal Dementia Caregivers
Brief Title: Effectiveness of an Online Training and Support Program (iSupport) for Informal Dementia Caregivers
Acronym: iSupportPT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: There were issues with the technical service provider of the platform iSupport-Portugal; the platform and its backoffice should be implemented by another service provider. A pilot study was conducted following the protocol of the full trial.
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: iSupport Portugal 208/18
Record Dates: First submitted 2019-09-19; First posted 2019-09-26 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Caregiver Subjective Burden; Depressive Symptoms; Anxiety Symptoms
Keywords: Informal caregivers; People with Dementia; Mental Health; Online training and support; Intervention Study
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Experimental parallel between-group design with two arms.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants are not unaware of the intervention received as they are active parts of the intervention. The data analyst will be blinded to the intervention assigned to the participants. Data collection at baseline and outcomes assessment are carried out in a computerized manner via study online platform and resorting to self-report/self-administered instruments, thus the researcher has no control or influence over the measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iSupport for dementia - European-Portuguese version (Experimental): Access, for 3 months, to an online self-help training and support program: iSupport for dementia - European-Portuguese version. The e-program offers information, skills training and support for informal caregivers of people with dementia. It comprises five modules, including twenty-three lessons on dementia and caregiver support. In line with good practices on digital engagement, the education plan can be personalized by the caregiver. This means that it can be adjusted to the person's availability and lessons can be selected according to particular needs. Each lesson includes interactive exercises with immediate feedback; and positive messages as well as 'skills certificates' are displayed when lessons are completed. Framed as a multi-component intervention, iSupport is grounded in problem-solving and cognitive behavioral therapy techniques including psycho-education, behavioral activation, cognitive reframing, relaxation and antecedent-behavior-consequence (ABC) analysis.
  Interventions: Behavioral: iSupport for dementia - European-Portuguese version
- Education-only e-book (Active Comparator): The control group will receive a minimal education-only intervention, consisting on an e-book. The manual contains information on relevant topics for dementia and caregiving, including basic information about dementia; practical tips on managing dementia; the changing needs of a person with dementia; dealing with care provision; caring for oneself (the caregiver) and finding emotional support; dealing with the death of the care receiver; relevant legislation (e.g. advance directives); how to get help; and how to reach the national Alzheimer's Association.
  Interventions: Other: e-book (comparator)

INTERVENTIONS:
Behavioral: iSupport for dementia - European-Portuguese version — iSupport for dementia, European-Portuguese version consists in an online self-help training and support program developed by the World Health Organization to to provide education, skills training and support to informal caregivers of people with dementia and culturally adapted to Portugal by the Institute of Biomedical Sciences Abel Salazar and CINTESIS. Framed as a multi-component intervention, iSupport is grounded in problem-solving and cognitive behavioral therapy techniques. The program comprises 23 lessons on dementia and caregiver support distributed by 5 modules: 'Introduction to dementia'; 'Being a carer'; 'Caring for me'; 'Providing everyday care' and 'Dealing with behavior changes'. The education plan can be personalized by the caregiver and each lesson includes interactive exercises with immediate feedback; and positive messages as well as 'skills certificates' are displayed when lessons are completed.
  Arms: iSupport for dementia - European-Portuguese version
Other: e-book (comparator) — The e-book contains information on relevant topics for dementia and caregiving, including basic information about dementia; practical tips on managing dementia; the changing needs of a person with dementia; dealing with care provision; caring for oneself (the caregiver) and finding emotional support; dealing with the death of the care receiver; relevant legislation (e.g. advance directives); how to get help; and how to reach the national Alzheimer's Association.
  Arms: Education-only e-book

SUMMARY:
Informal caregivers of people with dementia are at greater risk of developing physical and mental health problems when compared to the general population and to informal caregivers of people with other chronic diseases. Internet-based interventions have been explored in its potential to minimize the negative effects of caring, accounting for their ubiquitous nature, convenient delivery, potential scalability and presumed (cost)effectiveness. iSupport is a self-help online program developed by the World Health Organization to provide education, skills training and support to informal caregivers of people with dementia. This intervention study aims to determine the effectiveness of a Portuguese culturally adapted version of iSupport to decrease caregiver burden, symptoms of depression and anxiety, and to improve quality of life, positive aspects of caregiving and general self-efficacy. The study has two arms: access to "iSupport" for three months or access to an education-only e-book. iSupport is grounded in problem-solving and cognitive behavioral therapy techniques and it consists of 23 lessons organized around 5 modules: 'Introduction to dementia'; 'Being a carer', 'Caring for me', 'Providing everyday care', and 'Dealing with behaviour changes'.

One hundred and eighty four participants will be recruited by referral from national Alzheimer's associations. Participants will be included if they match the following criteria: being 18 years or older and provide e-consent; being a self-reported non-paid caregiver for at least 6 months; caring for a person with a formal diagnosis of Alzheimer's disease; being skilled to use internet; and experience a clinically relevant level of burden or depression or anxiety symptoms. Data is collected online, resorting to self-administered instruments, at baseline, 3 and 6 months after baseline. A two-sided alternative hypothesis was assumed for this study: Mean caregiver burden at 3 months after baseline is different in informal caregivers of people with dementia assigned to the iSupport program as in those assigned to a minimal education-only intervention. Findings from this intervention study will offer evidence to support an informed decision making on scaling up iSupport as a new intervention program with minimal costs aimed at minimizing the psychological distress of informal caregivers of people with dementia in Portugal and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Portuguese adults (≥18 years) (as self-reported and reported by professionals in the referral process);
* Giving consent to participate (Electronic Informed Consent);
* Providing non-paid care for at least 6 months at the time of the recruitment (as self-reported and reported by professionals in the referral process);
* Caring for a person holding a formal diagnosis of dementia (as reported by professionals in the referral process);
* Be skilled to use the internet (as self-reported and reported by professionals in the referral process);
* Experiencing either a clinically relevant level of subjective burden, as determined by a total score ≥ 21 on the Zarit Burden Interview or depression or anxiety symptoms, determined by a score ≥ 8 in at least one of the subscales of the Hospital Anxiety and Depression Scale.

Exclusion Criteria:

* Unable to comprehend written Portuguese (as reported by professionals in the referral process);
* Not having access to a device with internet connection at least twice a week (as self-reported and reported by professionals in the referral process);
* Declaring to care for a person in institutional care (e.g. nursing home or continued care unit) (as self-reported and reported by professionals in the referral process).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in subjective burden using the Zarit Burden Interview (ZBI) | Baseline, Month 3, Month 6
  Caregiver burden measured with the Zarit Burden Interview (ZBI), Portuguese validated version, total score. The instrument comprises 22 items answered on a 5-point scale, ranging from 0 (never) to 4 (almost always) except for the final question on global burden, rated from 0 (not at all) to 4 (extremely). Total score for the ZBI ranges from 0 to 88 points, with higher scores indicating greater burden. The ZBI has good internal consistency (0.89), test-retest and interrater reliability as well as construct and concurrent validity, including reports of positive correlation with depression symptoms and time devoted to care provision. Regarding the psychometric properties of ZBI in Portugal, face, content, ecological, discriminant and convergent validity were documented, along with test-retest reliability (ICC= 0.93, CI95% 0.88 - 0.96, p < 0.001) and internal consistency (α = 0.88). The ZBI is one of the most used instruments to measure burden in intervention studies with caregivers.

SECONDARY OUTCOMES:
Change from baseline in symptoms of depression and anxiety using the Hospital Anxiety and Depression Scale (HADS) | Baseline, Month 3, Month 6
  Symptoms of depression and anxiety measured through the Portuguese version of the Hospital Anxiety and Depression Scale (HADS), total scores. The instrument comprises two subscales with 7 items each, using a 4-point scale. Total scores for each scale range from 0 to 21, with higher scores indicating more severe anxiety or depression symptoms.
Change from baseline in quality of life using the WHOQOL-BREF | Baseline, Month 3, Month 6
  Quality of life measured by the Portuguese version of the WHOQOL-BREF Physical, Psychological, Social relationships and Environment, total transformed scores. The instrument contains 26 items, for total transformed scores ranging between 0 to 100 points, with higher scores denoting higher quality of life.
Change from baseline in Positive Aspects of Caregiving using the Positive Aspects of Caregiving (PAC) | Baseline, Month 3, Month 6
  Positive role appraisals mediating between the stressor and caregiver well-being, measured through the Portuguese version of Positive Aspects of Caregiving (PAC), total score. This instrument comprises 11 items answered in a 5-point scale, for a total score ranging between 11 to 55 points and higher scores representing more positive appraisals.
Change from baseline in General self-efficacy using the Generalized self-efficacy scale | Baseline, Month 3, Month 6
  General self-efficacy, measured through the total score of the Generalized self-efficacy scale. The scale comprises 10 items answered in a 4-point scale for a total score ranging between 10 to 40 points, and higher scores representing a higher general self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Soraia T Sousa, M.S., Principal Investigator — Instituto de Ciências Biomédicas Abel Salazar - Universidade do Porto; CINTESIS; Constança Paúl, PhD, Study Director — Instituto de Ciências Biomédicas Abel Salazar - Universidade do Porto; CINTESIS
Locations (1):
- Institute of Biomedical Sciences Abel Salazar, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teles S, Ferreira A, Paul C. Feasibility of an online training and support program for dementia carers: results from a mixed-methods pilot randomized controlled trial. BMC Geriatr. 2022 Mar 1;22(1):173. doi: 10.1186/s12877-022-02831-z. PMID 35232389
- [Derived] Teles S, Ferreira A, Seeher K, Freel S, Paul C. Online training and support program (iSupport) for informal dementia caregivers: protocol for an intervention study in Portugal. BMC Geriatr. 2020 Jan 8;20(1):10. doi: 10.1186/s12877-019-1364-z. PMID 31914936